CLINICAL TRIAL: NCT03705520
Title: Targeting Diet-Microbiome Interactions in the Pathogenesis of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: California Institute of Technology (Other); Purdue University (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Director, Division of Digestive Diseases, Rush University Medical Center
Other Study IDs: ORA 16111903
Record Dates: First submitted 2018-10-01; First posted 2018-10-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: PD; Parkinson's; Parkinson's Disease; Microbiome
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-Sectional: This cohort is composed of only medicated PD subjects and their spouse or 1st degree relative.
- Logitundinal: This cohort is composed of only non-medicated PD subjects and their spouse or first degree relative.

SUMMARY:
The purpose of this study is to evaluate the microbiome of medicated and non-medicated subjects diagnosed with Parkinson's disease. Where available, in comparison to the microbiome of a healthy spouse or 1st degree relative.

DETAILED DESCRIPTION:
First, a cross sectional study where the investigators will compare microbiome composition in subsets of PD and Multiple System Atrophy (MSA) patients whose household control agree to provide stool samples as well. Each household control subject will be evaluated to ensure there is no clinical evidence of neurological disorders including PD. Also, these subjects will complete a 24 hour diet recall questionnaire before stool collection and validated 3 month food frequency questionnaire to collect dietary information similar to PD patients. Each subject (including PD subjects) will complete a smell questionnaire and a sleep questionnaire to determine whether these "control" subjects have loss of smell or have REM sleep disorders because these conditions increase the risk of PD. For assessing smell, investigators will use the UPSIT questionnaire. For assessing REM sleep disorder, investigators will use RBD1Q which consists of a single question, answered "yes" or "no," as follows: "Has the subject ever been told, or suspected themselves that they seem to 'act out their dreams' while asleep (for example, punching, flailing their arms in the air, making running movements, etc.)?"

Second, in the longitudinal study, the investigators will collect stool every 3 months with 3 day diet questionnaire prior to each collection over 12 months and determine microbiome composition over time. Investigators will correlate the microbiome data with PD symptoms, diet and response to treatment and progression of disease. These studies will determine whether disease progression and factors such as PD medications and diet significantly impact microbiome composition. Furthermore, the investigators will determine whether changes in SCFA-producing bacteria and/or abnormal SCFA profiles correlate with severity of PD symptoms.

ELIGIBILITY:
Inclusion Criteria:

PD Subjects Inclusion:

* 40-80 years of age
* Previously diagnosed with Parkinson's disease
* Parkinson's disease stage between 1-4
* Are willing to participate in the study

Healthy control/ Spouse/ 1st degree relative Inclusion:

* Adults 40-80 years of age
* No clinical evidence of neurological disorders including Parkinson's disease
* Live in the same household as the Parkinson Disease patient or is a first degree relative of the PD patient or an independent healthy control
* Are willing to participate in the study

Exclusion Criteria:

PD Subjects Exclusion:

* History of GI diseases (except for hemorrhoids or occasional (<3 times a week) heartburn) like Inflammatory bowel disease or Celiac disease.
* Antibiotic use within last 12 weeks.
* Use of probiotic supplement except yogurt.
* Intentional change in diet.
* Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study. Low dose aspirin is allowed.

Healthy control/ Spouse/ 1st degree relative Exclusion:

* History of GI diseases (except for hemorrhoids or occasional (<3 times a week) heartburn) like Inflammatory bowel disease or Celiac disease.
* Antibiotic use within last 12 weeks.
* Use of probiotic supplement except yogurt.
* Intentional change in diet.
* Chronic use of NSAIDS. A washout period of 3 weeks is needed before the subject could be enrolled into the study. Low dose aspirin is allowed

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be selected from the neurology clinic, as well as a self-referrals.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Study microbiome composition to explain the exact nature of the dysbiosis (microbial imbalance) | 4 years
  The investigators anticipate confirming their prior findings that patients with PD have dysbiosis, and further identifying the nature of the dysbiosis including changes at the species and strain level.

SECONDARY OUTCOMES:
Identify the potential contributing factors for dysbiosis in PD | 4 years
  It is well established that environmental factors such as diet, as well as genetics, impact microbiome composition.Currently, there are no data for how environment impacts the microbiome in PD.
Determine how dysbiosis promotes PD | 4 years
  The investigators will determine SCFA (Short chain fatty acids) concentrations in serum and stool from early onset PD patients and healthy controls. The investigators will correlate serum, stool data, PD symptoms and disease severity obtained through validated PD questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, MD, Principal Investigator — Rush University Medical Center; Gian Pal, MD, Principal Investigator — Rush Univeristy Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No identifying information will be shared with other researchers.

DOCUMENTS (1):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT03705520/Prot_000.pdf